CLINICAL TRIAL: NCT05591924
Title: Prospective Observational Study of Biology of Critical Illness
Brief Title: Early Severe Illness TrAnslational BioLogy InformaticS in Humans
Acronym: ESTABLISH
Status: Recruiting | Type: Observational
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: London Health Sciences Centre (Other); Western University, Canada (Other); Western University (Other)
Responsible Party: Principal Investigator, Aleks Leligdowicz, Clinician Scientist, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Other Study IDs: 12145
Record Dates: First submitted 2022-10-05; First posted 2022-10-24 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-10

CONDITIONS: Sepsis; ARDS; Critical Illness; Neurocognitive Dysfunction; Shock, Septic; Ventilator Associated Pneumonia; Immune Suppression; Inflammation; SIRS
Keywords: Critical Care; Sepsis; ARDS; Inflammation; Immune responses; Neurocognition; Critical illness; Translational Biology
MeSH Terms: conditions — Sepsis; Critical Illness; Cognition Disorders; Shock, Septic; Pneumonia, Ventilator-Associated; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Biospecimen Retention: Samples With DNA — EDTA anticoagulated blood Heparin anticoagulated blood PAX gene tube Broncheoalveolar lavage fluid (BALF)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- ESTABLISH: Adults over 18 years of age admitted to the ICU within 48 hours and whose presentation to the Emergency Department was within 72h of ICU admission.
  Interventions: Procedure: Phelebotomy; Procedure: Broncheoalveolar Lavage; Procedure: Tracheal Aspirate; Procedure: Rectal Swab
- Healthy Controls: Adults over 18 years of age with no infectious symptoms, interaction with the health care system, or antimicrobial use in the past 14 days and no history of immunosuppression.
  Interventions: Procedure: Phelebotomy

INTERVENTIONS:
Procedure: Phelebotomy — Collection of 10mL of heparin anticoagulated blood, 10mL of EDTA anticoagulated blood, and 3mL of blood in a PAX gene tube
Procedure: Broncheoalveolar Lavage — Bronchioalveolar lavage fluid (BALF) samples will be obtained from participants who are mechanically ventilated, and a bronchoscopy is indicated as part of routine clinical care. The BALF will be collected by a qualified ICU physician using standard clinical practice. Briefly, patients will receive appropriate sedation and analgesia, a flexible video-bronchoscope will be inserted into the patient's airway, and bronchial segments will be identified. The bronchoscope will be wedged in the most appropriate lung segment and 40-100mL of sterile normal saline (NS) as clinically indicated, will be injected into the bronchoscope port with using a 50mL syringe. Next, the instilled NS (i.e.: lavage fluid) will be collected in a sterile container using gentle suction. The BALF will then be partitioned and sent to clinical laboratories, and the remaining BALF (10-20mL) will be used in the ESTABLISH research study.
  Groups: ESTABLISH
Procedure: Tracheal Aspirate — Tracheal Aspirate (TA) will be obtained from participants who have an endotracheal tube or a tracheostomy in situ at the time of ICU admission through out the ICU admission on the study days, as long as distal airway access is available.
  Groups: ESTABLISH
Procedure: Rectal Swab — A Rectal will be obtained at the time of ICU admission and on all study days during the ICU admission
  Groups: ESTABLISH

SUMMARY:
Advanced stages of the response to life-threatening infection, severe trauma, or other physiological insults often lead to exhaustion of the homeostatic mechanisms that sustain normal blood pressure and oxygenation. These syndromic presentations often meet the diagnostic criteria of sepsis and/or the acute respiratory distress syndrome (ARDS), the two most common syndromes encountered in the intensive care unit (ICU). Although critical illness syndromes, such as sepsis and ARDS, have separate clinical definitions, they often overlap clinically and share several common injury mechanisms. Moreover, there are no specific therapies for critically ill patients, and as a consequence, approximately 1 in 4 patients admitted to the ICU will not survive.

The purpose of this observational study is to identify early patient biologic factors that are present at the time of ICU admission that will help diagnose critical illness syndromes earlier, identify who could benefit most from specific therapies, and enable the discovery of new treatments for syndromes such as sepsis and ARDS.

DETAILED DESCRIPTION:
Background:

Critical illness syndromes, such as sepsis and ARDS, are associated with tremendous heterogeneity in patient predisposing risk factors, mechanisms of acute insult contributing to infection, presenting symptoms, response to therapies, as well as short and long-term outcomes. Since the first standardization of sepsis and ARDS definitions >30 years ago, significant insight into biological mechanisms contributing to critical illness syndromes have been made. However, there are many important unanswered questions that prevent accurate diagnosis, treatment, and prognosis of patients who present to the ICU with early symptoms consistent with critical illness.

Of the many gaps about the biology of sepsis and ARDS that remain unanswered, the following are particularly important: (1) what constitutes immune system dysregulation; (2) how the immune system response depends on interaction with the infecting pathogens; (3) what biologic traits distinguish other diagnoses that mimic these syndromes; (4) what are the mechanisms of genetic polymorphisms in patient outcomes. To address these questions and to improve our understanding of these complex and heterogenous syndromes, a multifaceted and collaborative approach is needed. This study will investigate the biology of early sepsis in critically ill patients by developing a longitudinal prospective observational cohort called Early Severe illness TrAnslational BioLogy InformaticS in Humans (ESTABLISH).

Specific objectives:

Objective 1: To study biologic mechanisms of immune system regulation during early critical illness. The main questions that will be addressed include: (1) how immune function at the time of admission and over the course of the ICU stay is related to clinical complications; (2) how anatomic compartmentalization of immune responses is associated with clinical complications; (3) how immune responses in different anatomic locations contribute to endothelial cell injury; (4) how macrophages contribute to distal organ injury and long-term clinical complications.

Objective 2: To characterize the host-pathogen interaction during early critical illness. The main question that will be addressed include: (1) how the microbial composition at the time of ICU admission affects the immune response; (2) how the change in host-pathogen interactions over time influence clinical complications.

Objective 3: To identify biologic traits that distinguish patients with early sepsis and ARDS from other critically ill patients. The main questions that will be addressed include: (1) are biological trains unique to sepsis and/or ARDS, or are they shared by other clinical diagnoses that mimic these syndromes?; (2) can accurately prognosticate clinically important short and long-term patient outcomes?; (3) are biologic traits associated with differential responses to therapies?

Objective 4: To study the molecular mechanisms of genetic polymorphisms associated with critical illness using induced pluripotent stem cells (iPSCs) derived from polymorphonuclear cells (PBMCs) from critically ill patients. The main questions that will be addressed include: (1) how do autologous iPSC-derived cell lineages interact with autologous plasma?; (2) how do iPSC-derived cell lineages respond to treatment with drugs related to genetic polymorphisms function?; (3) how do iPSC-derived lineages respond to treatment with drugs commonly used in the ICU?

Methods:

The ESTABLISH cohort will enroll patients within 48 hours of ICU admission who presented to the emergency department within 72 hours of ICU admission. Patients will be enrolled with deferred consent to enable the earliest possible collection of biological specimen. The biological specimen will include anticoagulated blood, a PAX gene tube, and a bronchioalveolar lavage fluid (BALF) sample (in mechanically ventilated patients, when bronchoscopy is clinically indicated) collected at the time of ICU admission (Day 0), and on 4 subsequent timepoints during the ICU admission (Days 1,3,7,14,21).

Data generated during ESTABLISH will be analyzed in batches on an ongoing, regular basis and will be objective-specific. Batch sample preparation and data analysis will minimize biological assay and methodological heterogeneity. Objective 1 and 2 data will be analyzed after enrollment of the first 50 patients, and every 50 patients after this. Objective 3 data will be analyzed after enrollment of the first 200 patients and every 200 patients after this.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old
* ≤48h since ICU admission
* ICU admission within 72h of presentation to the emergency department (ER)
* Clinical critical illness suspected on the basis of any one of the following:

  1. Altered mental status (GCS<15)
  2. Cardiovascular collapse (presence of any: Heart rate >90, systolic blood pressure <90, presence of vasopressors, lactate >2.0)
  3. Respiratory collapse (presence of any: respiratory rate >20, PaCO₂ <32 mm Hg, supplemental oxygen, invasive or non-invasive ventilation)
  4. Suspected severe infection (presence of any: temperature >38°C or <36°C, white blood cell (WBC) count >12,000/mm³ or <4,000/mm³, presence of 1 or more antibiotics at the time of ICU admission)

Exclusion Criteria:

* Age <18 years old
* >72h since ICU admission
* Admission to ICU in patients >72h after the presentation to the ER
* No evidence of critical illness (ICU admission due to bed-spacing)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Critically ill adults with early critical illness
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-04-26 (Actual); Primary Completion 2034-12-31 (Estimated); Study Completion 2034-12-31 (Estimated)

PRIMARY OUTCOMES:
Risk of developing nosocomial infections during ICU admission | Assessed daily until discharge from ICU, through study completion, an average of 1 year
  Development of any of the following: Ventilator Associated Pneumonia, Central Line Infections, Clostridium difficile-Associated Diarrhea, Blood stream infections
Severity of illness measured by APACHE score | At the time of ICU admission
  APACHE
Severity of illness measured by SOFA score | At the time of ICU admission
  SOFA
Severity of illness measured by MODS score | At the time of ICU admission
  MODS
Change in severity of illness measured by APACHE score | From the time of ICU admission, assessed daily until death or discharge from ICU, up to 12 months
  APACHE
Change in severity of illness measured by SOFA score | From the time of ICU admission, assessed daily until death or discharge from ICU, up to 12 months
  SOFA
Change in severity of illness measured by MODS score | From the time of ICU admission, assessed daily until death or discharge from ICU, up to 12 months
  MODS
Hospital disposition | Determined at the time of discharge from the hospital, through study completion, an average of 1 year
  Survival, death

SECONDARY OUTCOMES:
Neurocognitive dysfunction | 1, 6, and 12 months after ICU discharge
  Cambridge Brain Sciences (CBS) web-based neurocognitive battery
Physiological outcomes | 0, 24, 48, and 72 hours after ICU admission
  Ultrasound-identified volume responsiveness

CONTACTS AND LOCATIONS:
Overall Officials: Aleks Leligdowicz, MD PhD, Principal Investigator — Western University
Locations (1):
- Aleks Leligdowicz, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Biological specimen stored for future research may be eligible for collaborative future studies. Collaborators will be required to complete a study plan and be approved by the Lawson ethics board and/or the Western University HSREB.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Access Criteria: Collaborating researchers must be approved by the Lawson ethics board and/or the Western University HSREB.

REFERENCES:
- [Background] Micic S, Illic V, Isvaneski M. Correlation of hormone and histologic parameters in infertile men with varicocele. Urol Int. 1983;38(3):187-90. doi: 10.1159/000280888. PMID 6408778
- [Background] Maslove DM, Tang B, Shankar-Hari M, Lawler PR, Angus DC, Baillie JK, Baron RM, Bauer M, Buchman TG, Calfee CS, Dos Santos CC, Giamarellos-Bourboulis EJ, Gordon AC, Kellum JA, Knight JC, Leligdowicz A, McAuley DF, McLean AS, Menon DK, Meyer NJ, Moldawer LL, Reddy K, Reilly JP, Russell JA, Sevransky JE, Seymour CW, Shapiro NI, Singer M, Summers C, Sweeney TE, Thompson BT, van der Poll T, Venkatesh B, Walley KR, Walsh TS, Ware LB, Wong HR, Zador ZE, Marshall JC. Redefining critical illness. Nat Med. 2022 Jun;28(6):1141-1148. doi: 10.1038/s41591-022-01843-x. Epub 2022 Jun 17. PMID 35715504
- [Background] Jung RT. Obesity as a disease. Br Med Bull. 1997;53(2):307-21. doi: 10.1093/oxfordjournals.bmb.a011615. PMID 9246838
- [Background] Yacubian EM, Rosemberg S, Marie SK, Valerio RM, Jorge CL, Cukiert A. Double pathology in Rasmussen's encephalitis: etiologic considerations. Epilepsia. 1996 May;37(5):495-500. doi: 10.1111/j.1528-1157.1996.tb00597.x. PMID 8617180
- [Background] Tandon SP, Mishra MM. Effect of sodium, manganese and zinc on the activity of nitrobacter agilis. Zentralbl Bakteriol Parasitenkd Infektionskr Hyg. 1969;123(4):399-402. No abstract available. PMID 5395141
- [Background] Yoshino M, Murakami K. The regulatory role of spermine and fatty acid in the interaction of AMP deaminase with phosphofructokinase. Biochim Biophys Acta. 1982 Dec 17;719(3):474-9. doi: 10.1016/0304-4165(82)90235-5. PMID 6295506
- [Background] Aono R. Improvement of organic solvent tolerance level of Escherichia coli by overexpression of stress-responsive genes. Extremophiles. 1998 Aug;2(3):239-48. doi: 10.1007/s007920050066. PMID 9783171
- [Background] Kaplan A, Matsue H, Shibaki A, Kawashima T, Kobayashi H, Ohkawara A. The effects of cyclosporin A and FK506 on proliferation and IL-8 production of cultured human keratinocytes. J Dermatol Sci. 1995 Sep;10(2):130-8. doi: 10.1016/0923-1811(95)00395-9. PMID 8534611
- Available data/document: C3RP Laboratory Website — https://c3rp.org/leligdowiczlab